CLINICAL TRIAL: NCT04275947
Title: The COVID-19 Mobile Health Study, a Large-scale Clinical Observational Study Using nCapp
Brief Title: The COVID-19 Mobile Health Study (CMHS)
Acronym: CMHS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Alliance Against Lung Cancer (Other)
Collaborators: Shanghai Respiratory Research Institution (Unknown)
Responsible Party: Principal Investigator, Bai Chunxue, Chair, Chinese Alliance Against Lung Cancer
Other Study IDs: CAALC-008-CMHS
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training
  Interventions: Other: nCapp, a cell phone-based auto-diagnosis system
- Validation
  Interventions: Other: nCapp, a cell phone-based auto-diagnosis system

INTERVENTIONS:
Other: nCapp, a cell phone-based auto-diagnosis system — Combined with 15 questions online, and a predicated formula to auto-diagnosis of the risk of COVID-19

SUMMARY:
This study evaluates a brand-new cell phone-based auto-diagnosis system, which is based on the clinical guidelines, clinical experience, and statistic training model. We will achieve secure and 1st hand data from physicians in Wuhan, which including 150 cases in the training cohort and 300 cases in the validation cohort.

ELIGIBILITY:
Inclusion Criteria:

* High risk of COVID-19
* RT-PCR test result of SAR2-CoV-19

Exclusion Criteria:

* Not available for RT-PCR test result of SAR2-CoV-19

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: -High risk of COVID-19
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of nCapp COVID-19 risk diagnostic model | 1 day
  Sensitivity, specificity and area under the ROC curve of nCapp model

CONTACTS AND LOCATIONS:
Overall Officials: Chunxue Bai, Principal Investigator — Shanghai Respiratory Research Institution
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
The anonymous clinical data for training and validation the model

REFERENCES:
- [Background] Yang D, Zhang X, Powell CA, Ni J, Wang B, Zhang J, Zhang Y, Wang L, Xu Z, Zhang L, Wu G, Song Y, Tian W, Hu JA, Zhang Y, Hu J, Hong Q, Song Y, Zhou J, Bai C. Probability of cancer in high-risk patients predicted by the protein-based lung cancer biomarker panel in China: LCBP study. Cancer. 2018 Jan 15;124(2):262-270. doi: 10.1002/cncr.31020. Epub 2017 Sep 20. PMID 28940455